CLINICAL TRIAL: NCT03690336
Title: Adverse Event Data Collection From External Registries on Nonacog Beta Pegol
Status: Enrolling by invitation | Type: Observational
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Other Study IDs: NN7999-4413; U1111-1212-4050 (Other: World Health Organization (WHO)); EUPAS25696 (Registry Identifier: EU PAS Register)
Record Dates: First submitted 2018-09-21; First posted 2018-10-01 (Actual); Last update posted 2025-06-02 (Actual); Status verified 2025-05

CONDITIONS: Haemophilia B
MeSH Terms: conditions — Hemophilia B | interventions — nonacog beta pegol

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with haemophilia B: Patients with haemophilia B treated with nonacog beta pegol who report adverse events to the PedNet and EUHASS, and possibly other national or international registries.
  Interventions: Drug: Nonacog beta pegol

INTERVENTIONS:
Drug: Nonacog beta pegol — Treatment with commercially available nonacog beta pegol according to routine clinical practice at the discretion of the treating physician.

SUMMARY:
The purpose of this study is to collect data on adverse events from third party registries that include information about adverse events from patients with haemophilia B treated with nonacog beta pegol. The third party registries include PedNet Haemophilia Registry (PedNet) and the European Haemophilia Safety Surveillance System (EUHASS). Data from national and international registries in countries where nonacog beta pegol has been approved and marketed could be included in the data collection.

ELIGIBILITY:
Inclusion Criteria:

- Participation in the PedNet Registry and/or the European Haemophilia Safety Surveillance System (EUHASS), or other national and international registries

Exclusion Criteria:

- Not applicable as this is a study collecting third-party data from registries

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with haemophilia B
Sampling Method: Non-Probability Sample
Enrollment: 10 (Estimated)
Dates: Start 2018-10-01 (Actual); Primary Completion 2027-10-01 (Estimated); Study Completion 2027-10-01 (Estimated)

PRIMARY OUTCOMES:
Adverse Drug Reactions (ADRs) reported to the registries with suspected relation to nonacog beta pegol in patients with haemophilia B | From start of data collection (week 0) to end of data collection (after 9 years)
  Number of events (renal, hepatic, neurodevelopmental, neurocognitive, neurologic or psychiatric events)

SECONDARY OUTCOMES:
Other ADRs reported to the registries during the study period with suspected relation to nonacog beta pegol in patients with haemophilia B | From start of data collection (week 0) to end of data collection (after 9 years)
  Number of events (de novo FIX inhibitors more than or equal to 0.6 Bethesda units); anaphylaxis and other allergic reactions; thromboembolic events)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Transparency (2834), Study Director — Novo Nordisk A/S
Locations (2):
- PedNet Haemophilia Registry, Baarn, Netherlands
- European Haemophilia Safety Surveillance Registry, Sheffield, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
According to the Novo Nordisk disclosure commitment on novonordisk-trials.com
URL: http://novonordisk-trials.com